CLINICAL TRIAL: NCT05287204
Title: Critical Illness Myopathy and Trajectory of Recovery in Acute Kidney Injury (AKI) Requiring Continuous Renal Replacement Therapy (CRRT): A Prospective Observational Trial
Brief Title: Critical Illness Myopathy and Trajectory of Recovery in AKI Requiring CRRT
Status: Active, not recruiting | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Benjamin Griffin, Assistant Professor, University of Iowa
Other Study IDs: 202002328
Record Dates: First submitted 2021-10-20; First posted 2022-03-18 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury; Critical Illness Myopathy; Dialysis; Complications
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples and effluent samples will be stored for metabolomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI-RRT: Adults admitted to the ICU with AKI requiring CRRT with study enrollment within 48 hours of CRRT initiation.
  Interventions: Diagnostic Test: Musculoskeletal ultrasound; Diagnostic Test: Assessments of muscle strength and physical function; Diagnostic Test: Metabolomics
- Historical Controls: The controls for the ICU phase will be 41 critically ill adults without AKI-RRT in whom similar measurements of muscle size, quality, and function were collected in a recent prior study [PubMed ID: 33148301]. The controls for the recovery phase will come from an ongoing prospective observational study being performed at the University of Kentucky, which will include outpatient functional assessments performed on 200 ICU survivors (NCT05537298).
  Interventions: Diagnostic Test: Musculoskeletal ultrasound; Diagnostic Test: Assessments of muscle strength and physical function

INTERVENTIONS:
Diagnostic Test: Musculoskeletal ultrasound — Ultrasound of rectus femoris to determine cross-sectional area, muscle thickness, echo intensity.
Diagnostic Test: Assessments of muscle strength and physical function — A battery of tests of physical function and muscle strength (see outcomes section for details).
Diagnostic Test: Metabolomics — Using metabolomic analysis, concentrations of amino acids and other important analytes will be measured in patient plasma and CRRT effluent
  Groups: AKI-RRT

SUMMARY:
The purpose of this study is to determine whether patients with acute kidney injury requiring renal replacement therapy have a higher incidence of muscle wasting than controls and whether the course of recovery is longer compared to controls.

DETAILED DESCRIPTION:
Acute kidney injury (AKI), the abrupt loss of kidney function, is a common complication that affects more than half of all intensive care unit (ICU) admissions, and it is associated with substantially higher rates of morbidity and mortality in both the short- and the long-term. This is especially true in patients with AKI requiring renal replacement therapy (AKI-RRT), also known as dialysis. An understudied mechanism by which AKI-RRT may contribute to poor clinical outcomes, both in the hospital and after discharge, is through its impact on muscle mass and muscle function. AKI of any severity is known to alter tissue utilization of amino acids, and preliminary data suggest that RRT in the ICU may exacerbate muscle dysfunction through the removal of large quantities of amino acids from the patient's plasma. This study will determine whether patients with AKI-RRT have greater lean muscle loss over 1 week than historical critically ill controls, whether patients with AKI-RRT have diminished recovery of muscle mass and function at 1-3 months following discharge compared to controls, and whether changes in plasma levels of amino acids during hospitalization correlate with loss of muscle function or lack of recovery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* AKI requiring CRRT, with enrollment within 48 hours of CRRT initiation

Exclusion Criteria:

* ICU admission for >7 days
* RRT of any kind at any time prior to ICU admission
* Chronic kidney disease (CKD) with estimated glomerular filtration rate <20 mL/min/1.73 m2 as calculated by the 2021 CKD-EPI equation
* underlying muscle disorders or muscle atrophy such as quadriplegia or hemiplegia, stroke with residual motor deficits, end-stage liver disease, active alcohol use disorder, active malignancy (other than non-melanoma skin cancer) within 1 year, burns, or other baseline neuromuscular disease
* pregnancy
* concomitant use of other extracorporeal support devices such as ventricular assist devices or extracorporeal membrane oxygenation
* anticipated inability to engage in weight-bearing testing after discharge (e.g., trauma or orthopedic surgery)
* subjects will be ineligible for outpatient testing if they remain on RRT in the week prior to the research appointment

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of critically ill patients with acute kidney injury requiring continuous renal replacement therapy in an ICU setting.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
ICU Stage: rectus femoris (RF) cross-sectional area (CSA) | 7 days
  RF CSA as assessed by musculoskeletal ultrasound (MSKUS) will be measured at day 0 (study enrollment within 48 hours of CRRT initiation), at day 3, and at day 7 (or at ICU discharge if before day 7).
ICU Stage: RF muscle thickness (mT) | 7 days
  RF mT as assessed by MSKUS will be measured at day 0 (study enrollment within 48 hours of CRRT initiation), at day 3, and at day 7 (or at ICU discharge if before day 7).
ICU Stage: RF echo intensity (EI) | 7 days
  RF EI as assessed by MSKUS will be measured at day 0 (study enrollment within 48 hours of CRRT initiation), at day 3, and at day 7 (or at ICU discharge if before day 7).
RF CSA at discharge | 1 month
  RF CSA as assessed by MSKUS will be measured at hospital discharge.
RF mT at discharge | 1 month
  RF mT as assessed by MSKUS will be measured at hospital discharge.
RF EI at discharge | 1 month
  RF EI as assessed by MSKUS will be measured at hospital discharge.
RF CSA at post-discharge outpatient visit | 1-3 months
  RF CSA as assessed by MSKUS will be measured at outpatient follow-up visit.
RF mT at post-discharge outpatient visit | 1-3 months
  RF mT as assessed by MSKUS will be measured at outpatient follow-up visit.
RF EI at post-discharge outpatient visit | 1-3 months
  RF mT as assessed by MSKUS will be measured at outpatient follow-up visit.
ICU Stage: ICU Mobility Scale | 7 days
  The ICU Mobility Scale is an 11-point scale ranging from 0-10 which involves scoring a patient's maximum level of mobility in the prior 24-hour period. The ICU Mobility Scale will be performed at the same 3 time points as the MSKUS assessments.
Muscle Strength - Medical Research Council Sum-score (MRC-ss) at discharge | 1 month
  MRC-ss is a measure of global peripheral muscle strength that is the current clinical standard for diagnosing ICU-acquired weakness. Muscle strength is assessed by physical exam and rated on an ordinal scale (0-5) at six bilateral muscle groups: shoulder abductors, elbow flexors, wrist extensors, hip flexors, knee extensors, and ankle dorsiflexors.
Muscle Strength - MRC-ss at post-discharge outpatient visit | 1-3 months
  MRC-ss is a measure of global peripheral muscle strength that is the current clinical standard for diagnosing ICU-acquired weakness. Muscle strength is assessed by physical exam and rated on an ordinal scale (0-5) at six bilateral muscle groups: shoulder abductors, elbow flexors, wrist extensors, hip flexors, knee extensors, and ankle dorsiflexors.
Muscle Strength - knee extension by hand-held dynamometry (HHD) at hospital discharge | 1 month
  Maximal isometric knee extensor muscle strength as measured by HHD.
Muscle Strength - knee extension by HHD at post-discharge outpatient visit | 1-3 months
  Maximal isometric knee extensor muscle strength as measured by HHD.
Muscle Strength - Grip Strength at hospital discharge | 1 month
  Maximal isometric grip strength as measured by hand-grip dynamometry (HGD)
Muscle Strength - Grip Strength at post-discharge outpatient visit | 1-3 months
  Maximal isometric grip strength as measured by HGD
Physical Function - Short Physical Performance Battery (SPPB) at discharge | 1 month
  SPPB is a performance-based composite test with a total of 12 points including components of balance (side-by-side stand, semi-tandem stand, and full-tandem stand), chair-to-stand test, and 4-meter habitual gait speed used to assess physical function and physical frailty.
Physical Function - SPPB at post-discharge outpatient visit | 1-3 months
  SPPB is a performance-based composite test with a total of 12 points including components of balance (side-by-side stand, semi-tandem stand, and full-tandem stand), chair-to-stand test, and 4-meter habitual gait speed used to assess physical function and physical frailty.
TUG Test at post-discharge outpatient visit | 1-3 months
  The Timed Up and Go (TUG) test assesses the time (in seconds) for a subject to stand on command from a seated position, walk 3 meters, turn around, walk back to the chair, and sit down, thereby assessing mobility, physical function, and fall risk.
Physical Function - 6-minute walk test (6MWT) at post-discharge outpatient visit | 1-3 months
  The 6MWT assesses the distance a subject can walk in six minutes, providing a global representation of physical function and cardiopulmonary endurance.
Quality of Life testing using EuroQol Group 5-dimension 5-level (EQ-5D-5L) questionnaire at post-discharge outpatient visit | 1-3 months
  The EQ-5D-5L is a standardized measure of health status developed by the Euro-Qol Group to provide an assessment of health for clinical and economic appraisal.
Physical Function - Clinical Frailty Scale (CFS) at post-discharge outpatient visit | 1-3 months
  CFS is a widely adopted judgement-based tool to screen for frailty and to broadly stratify degrees of fitness and frailty.
Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Questionnaire at post-discharge outpatient visit | 1-3 months
  The FACIT-F scale is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function.
36-Item Short Form Health Survey Physical Function Scale (SF-36) at post-discharge outpatient visit | 1-3 months
  The SF-36 is a 36-item patient-reported survey of health commonly used to evaluate adult patients which contains 8 domains, including a physical function scale based on 10 of the 36 items which has been shown to have high reliability.
Return to driving | 1-3 months
  Yes / No outcome assessed at the outpatient follow-up visit
Return to work or hobby | 1-3 months
  Yes / No outcome assessed at the outpatient follow-up visit
Hospital Readmission | 1-3 months
  Yes / No outcome assessed at the outpatient follow-up visit
Emergency Department Visit | 1-3 months
  Yes / No outcome assessed at the outpatient follow-up visit

SECONDARY OUTCOMES:
ICU Stage: Changes in Plasma Metabolome | 7 days
  Plasma samples will be obtained at day 0 (study enrollment within 48 hours of CRRT initiation), at day 3, and at day 7 (or at ICU discharge if before day 7) and metabolomic analysis will be performed to determine if changes in the plasma metabolome with CRRT initiation correlate with parameters of muscle wasting and/or trajectory of recovery of muscle weakness.
ICU Stage: Changes in CRRT Effluent Metabolome | 7 days
  CRRT effluent samples will be obtained at day 0 (study enrollment within 48 hours of CRRT initiation), at day 3, and at day 7 (or at ICU discharge if before day 7) and metabolomic analysis will be performed to determine if changes in the effluent metabolome with CRRT initiation correlate with parameters of muscle wasting and/or trajectory of recovery of muscle weakness.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - University of New Mexico, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Teixeira JP, Mayer KP, Griffin BR, George N, Jenkins N, Pal CA, Gonzalez-Seguel F, Neyra JA. Intensive Care Unit-Acquired Weakness in Patients With Acute Kidney Injury: A Contemporary Review. Am J Kidney Dis. 2023 Mar;81(3):336-351. doi: 10.1053/j.ajkd.2022.08.028. Epub 2022 Nov 2. PMID 36332719
- [Background] Mayer KP, Thompson Bastin ML, Montgomery-Yates AA, Pastva AM, Dupont-Versteegden EE, Parry SM, Morris PE. Acute skeletal muscle wasting and dysfunction predict physical disability at hospital discharge in patients with critical illness. Crit Care. 2020 Nov 4;24(1):637. doi: 10.1186/s13054-020-03355-x. PMID 33148301
- [Background] Mayer KP, Welle MM, Evans CG, Greenhill BG, Montgomery-Yates AA, Dupont-Versteegden EE, Morris PE, Parry SM. Muscle Power is Related to Physical Function in Patients Surviving Acute Respiratory Failure: A Prospective Observational Study. Am J Med Sci. 2021 Mar;361(3):310-318. doi: 10.1016/j.amjms.2020.09.018. Epub 2020 Oct 3. PMID 33189316
- [Background] Mayer KP, Dhar S, Cassity E, Denham A, England J, Morris PE, Dupont-Versteegden EE. Interrater Reliability of Muscle Ultrasonography Image Acquisition by Physical Therapists in Patients Who Have or Who Survived Critical Illness. Phys Ther. 2020 Aug 31;100(9):1701-1711. doi: 10.1093/ptj/pzaa068. PMID 32302406
- [Background] Mayer KP, Ortiz-Soriano VM, Kalantar A, Lambert J, Morris PE, Neyra JA. Acute kidney injury contributes to worse physical and quality of life outcomes in survivors of critical illness. BMC Nephrol. 2022 Apr 7;23(1):137. doi: 10.1186/s12882-022-02749-z. PMID 35392844
- [Derived] Mayer KP, Teixeira JP, Gonzalez-Seguel F, Tran VQ, Gross JM, Horikawa-Strakovsky A, Pal CA, Shareef ZT, Puffer Israel H, Wen Y, Griffin BR, Neyra JA. Acute skeletal muscle wasting in patients with acute kidney injury requiring continuous kidney replacement therapy: A prospective multicenter study. J Crit Care. 2025 Oct;89:155142. doi: 10.1016/j.jcrc.2025.155142. Epub 2025 Jun 12. PMID 40513259
- [Derived] Gonzalez-Seguel F, Tran VQ, Pal CA, Shareef ZT, Israel HP, Horikawa-Strakovsky A, Wen Y, Griffin BR, Neyra JA, Teixeira JP, Mayer KP. Inter-rater reliability of muscle ultrasonography performed by multidisciplinary novice sonographers in the evaluation of critically ill patients with acute kidney injury requiring continuous kidney replacement therapy. Ren Fail. 2025 Dec;47(1):2472990. doi: 10.1080/0886022X.2025.2472990. Epub 2025 Mar 11. PMID 40069097
- [Derived] Teixeira JP, Griffin BR, Pal CA, Gonzalez-Seguel F, Jenkins N, Jones BM, Yoshida Y, George N, Israel HP, Ghazi L, Neyra JA, Mayer KP. Critical illness myopathy and trajectory of recovery in acute kidney injury requiring continuous renal replacement therapy: a prospective observational trial protocol. BMJ Open. 2023 May 22;13(5):e072448. doi: 10.1136/bmjopen-2023-072448. PMID 37217272

DOCUMENTS (2):
  • Study Protocol (2023-01-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT05287204/Prot_000.pdf
  • Informed Consent Form (2023-01-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT05287204/ICF_001.pdf